CLINICAL TRIAL: NCT03819010
Title: Neoadjuvant Letrozole + Palbociclib in Patients With II-IIIB BC,HR+, HER2-, Phenotype and Pretreatment Recurrence Score(RS):18-25 or 26-100 by Oncotype DX Breast RS Assay.Analysis of RS and Pathological Changes at Surgery
Brief Title: Neoadjuvant Letrozole and Palbociclib in Patients With Stage II-IIIB Breast Cancer, HR+, HER2 -
Acronym: DxCARTES
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MedSIR (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MedOPP199; 2018-001702-28 (EudraCT Number)
Record Dates: First submitted 2019-01-04; First posted 2019-01-28 (Actual); Last update posted 2020-11-27 (Actual); Status verified 2019-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — palbociclib

STUDY DESIGN:
Intervention Model Description: This is an international, multicenter, open-label, non-comparative, Simon´s two-stage design, phase II clinical trial.
Masking Description: Two arms of patients (according to Recurrence Score results), but both arms will be treated with the same treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pre treatment Recurrence Score:18-25 Letrozole + Palbociclib (Active Comparator): Letrozole (2,5 mg/day during 28 days of each Cycle) + Palbociclib (125mg/day during 21 days of each cycle of 28 days) as neoadjuvant treatment during 6 cycles before surgery of Breast Cancer interventions: Letrozol (2,5 mg/day during 28 days of each Cycle)+ Palbociclib(125mg/day during 21 days of each cycle of 28 days) as neoadjuvant treatment during 6 cycles before surgery of Breast Cancer
  Interventions: Drug: Pre treatment Recurrence Score:18-25 Letrozole + Palbociclib
- Pre treatment Recurrence Score:26-100 Letrozole + Palbociclib (Active Comparator): Letrozole (2,5 mg/day during 28 days of each Cycle) + Palbociclib (125mg/day during 21 days of each cycle of 28 days) as neoadjuvant treatment during 6 cycles before surgery of Breast Cancer interventions: Letrozol (2,5 mg/day during 28 days of each Cycle)+ Palbociclib(125mg/day during 21 days of each cycle of 28 days) as neoadjuvant treatment during 6 cycles before surgery of Breast Cancer
  Interventions: Drug: Pre treatment Recurrence Score:26-100 Letrozole + Palbociclib

INTERVENTIONS:
Drug: Pre treatment Recurrence Score:18-25 Letrozole + Palbociclib — Letrozole(2,5 mg/day during 28 days of each Cycle) + Palbociclib(125mg/day during 21 days of each cycle of 28 days) as neoadjuvant treatment during 6 cycles before surgery of Breast Cancer for patients with pre-treatment recurrence Score of 18-25
  Other Names: None othe intervention name
  Arms: Pre treatment Recurrence Score:18-25 Letrozole + Palbociclib
Drug: Pre treatment Recurrence Score:26-100 Letrozole + Palbociclib — Letrozole(2,5 mg/day during 28 days of each Cycle) + Palbociclib(125mg/day during 21 days of each cycle of 28 days) as neoadjuvant treatment during 6 cycles before surgery of Breast Cancer for patients with pre-treatment recurrence Score of 26-100
  Other Names: None othe intervention name
  Arms: Pre treatment Recurrence Score:26-100 Letrozole + Palbociclib

SUMMARY:
This is an international, multicenter, open-label, non-comparative, Simon´s two-stage design, phase II clinical trial.

DETAILED DESCRIPTION:
Primary objective:

To explore after 6 months of treatment the ability of palbociclib in combination with letrozole to induce global molecular changes measured by either the Oncotype DX Breast Recurrence Score® (the "Assay") test result at surgery (post-treatment Recurrence Score® (RS) result), or pathological Complete Response (pCR) in patients with aggressive luminal tumors (pre-treatment RS result 18-25 or 26-100, and Ki67≥ 20).

Secondary objectives:

BIOLOGY

* To explore the ability of palbociclib in combination with letrozole to induce global molecular changes measured by post-treatment RS result, in patients with aggressive luminal tumors (pre-treatment RS result 18-25 and Ki67≥ 20) after 6 months of treatment.
* To explore the ability of palbociclib in combination with letrozole to induce global molecular reduction measured by either the post-treatment RS result, and/or Residual Cancer Burden (RCB), and/or Ki67 in patients with aggressive luminal tumors (pre-treatment RS result 18-25 or 26-100 and Ki67 ≥ 20) after 6 months of treatment.
* To verify the ability of palbociclib in combination with letrozole to induce global molecular reduction (measured as either post-treatment RS≤25 or RCB score of 0-I) in >35% of patients in cohort B with pre-treatment RS 26-100;
* To verify the ability of palbociclib in combination with letrozole to induce increase in RS result (measured as post-treatment RS 26-100) in <3% of patients in cohort A with pre-treatment RS 18-25;
* To evaluate the concordance rate between the RCB score (0- I vs. II-III) and the post-treatment RS result in both cohorts of patients after treatment with palbociclib in combination with letrozole;
* To evaluate the concordance rate between the preoperative endocrine prognostic index (PEPI) score and post-treatment RS result in both cohorts of patients after treatment with palbociclib in combination with letrozole;
* To evaluate the concordance rate between the pCR and the post-treatment RS result in both cohorts of patients after treatment with palbociclib in combination with letrozole;
* To determine the change in RS result as measured by median absolute value or median percentage after 6 months of treatment: from pre-treatment RS 18-25 to post-treatment RS 0-17 for patients in cohort A and from pre-treatment RS 26-100 to post-treatment RS≤25 for patients in cohort B.

EFFICACY

* To determine the Overall Response Rate (ORR) of patients treated with palbociclib in combination with letrozole.
* To evaluate the Maximum Tumor Shrinkage of palbociclib in combination with letrozole.
* To determine the rate of breast conserving surgery.

SAFETY

• To assess the safety and tolerability of palbociclib in combination with letrozole.

A two-stage Simon's statistical design will be used for both cohorts (minimax design in co-hort B and optimal design in cohort A). A total of 66 patients will be enrolled into this trial, N=33 patients in cohort with high-risk tumors (Cohort B: pre-treatment RS>25) and N=33 patients in cohort with intermediate-risk tumors (Cohort A: pre-treatment RS18-25).

The accrual goal will be of 26 patients (N=13 patients in each cohort) during the first stage. The interim analysis has been planned after 15 patients (cohort B) and 9 patients (cohort A) will be available for biological response evaluation, and in case of positive findings, the trial will recruit additional 40 patients (N=20 patients in each cohort).

* The study would be defined as positive at final analysis in the cohort B (pre-treatment RS>25), if 8 or more than 8 patients with biological signal (post-treatment RS≤25) are observed (≥28.6%) among 28 evaluable patients.
* The study would be defined as positive at final analysis in the cohort A (pre-treatment RS18-25), if 25 or more than 25 patients with biological stabilization (post-treatment RS≤25) are observed (≥89.3%) among 28 evaluable patients.

Study treatment management

After signing the informed consent form (ICF) and confirmed pre- eligibility, patients will be pre-registered in the study. A tissue biopsy from the primary breast cancer has to be provided at screening and will be used to perform central confirmation of Ki67 levels and HR status, as well as central assessment of RS. Pre-registered patients can receive up to 4 weeks of letrozole before inclusion; pre-menopausal patients will require to combine it with a Luteinizing Hormone-Releasing Hormone (LHRH) analogue. Patients are eligible to enter one of the two cohorts according to RS assessment as follow:

* Cohort A: patients with pre-treatment RS 18-25;
* Cohort B: patients with pre-treatment RS 26-100. Patients with pre-treatment RS 0-17 will be considered not eligible. Patients allocated to the cohort A or B will receive 24 weeks of palbociclib (for 21 days every 4 weeks) in combination with letrozole (once daily, beginning on day 1 and continuing through day 28 of every 28-day cycle). Premenopausal women must also be treated with an LHRH analogue during the treatment phase.

ELIGIBILITY:
IInclusion criteria

Patients must meet ALL of the following inclusion criteria to be eligible for enrolment into the study:

1. Female patients over 18 years of age.
2. Patients have been informed about the nature of study, have agreed to participate in the study, and have signed the informed consent form prior to participation in any study-related activities.
3. Premenopausal and postmenopausal women. Premenopausal women must be treated with LHRH analogue since patient pre- registration. Premenopausal or postmenopausal status should have been established before starting study treatment with letrozole plus palbociclib based on the following classification:

   1. Postmenopausal status is defined as either:

      * Prior bilateral oophorectomy; Or
      * Age>60 years; Or
      * Age<60 years and amenorrhoeic for 12 months in the absence of chemotherapy, tamoxifen, toremifene or ovarian suppression, and follicle-stimulating hormone (FSH) and estradiol in postmenopausal range.
   2. Premenopausal status is defined as all those women who do not meet any of above criteria.
4. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1.
5. Histologically confirmed infiltrating breast cancer.
6. HR-positive (estrogen receptor [ER]-positive and/or progesterone receptor [PgR]-positive) EBCs (breast cancers that have at least 10% of cells staging positive for ER and/or PgR). ER and/or PgR status will be centrally confirmed by using immunohistochemistry (IHC) testing for an Allred score of 6-8 in at least one of them.
7. Patients with HER2-negative breast cancer through in situ hybridization test (fluorescence in situ hybridization [FISH], chromogenic in situ hybridization [CISH], or silver enhanced in situ hybridization [SISH]) or negative immunohistochemical status of 0, 1+, or 2+. If IHC is 2+, a negative in situ hybridization (FISH, CISH, or SISH) test is required.
8. Ki67 levels ≥ 20% confirmed by IHC testing in a central laboratory.
9. Tumor size > 2,0 cm (T2-4 according to TNM staging system, but always > 2,0 cm) by mammogram, breast ultrasound, or breast magnetic resonance imaging (MRI).
10. Patients must have a measurable disease by mammogram and/or breast ultrasound.
11. Patients with two significant lesions (both larger than 1 cm and with more than 1 cm distance between them) will require tumor sample from both lesions and proper preoperative marking of both. To be registered, both lesions should fulfil inclusion criteria 5 and 6 and both tumor samples will be submitted. Patient with more than 2 significant lesions will not be eligible.
12. Limited node involvement (N0-2, according to TNM staging system), assessed by ultrasound. Sentinel lymph node biopsy or axillary dissection, are allowed.
13. No metastatic disease (M0, according to TNM staging system).
14. Available pre-treatment tissue sample (biopsy) material (formalin- fixed paraffin-embedded (FFPE) for central confirmation and RS evaluation by the Assay.
15. Patients agree to collection of tissue biopsy from the primary breast cancer at the time of study inclusion (screening), at Cycle 1 Day 14 of treatment, and after 24 weeks (surgery), or if experience intolerable side effects, disease progression, or withdraw during 24 weeks of study treatment.
16. No prior chemotherapy, endocrine, or radiation therapy for current disease.
17. Adequate organ function:

    1. Hematological: White blood cell (WBC) count ≥ 3.0 x 109/L, absolute neutrophil count (ANC) ≥ 1.5x 109/L, platelet count ≥ 75.0 x109/L, and hemoglobin ≥ 10.0 g/dL (≥ 6.2 mmol/L).
    2. Hepatic: Bilirubin ≤ 1.5 times the upper limit of normal (x ULN) (or total bilirubin ≤ 3.0 x ULN or direct bilirubin ≤ 1.5 x ULN in patients with well-documented Gilbert's syndrome); alkaline phosphatase (ALP) ≤ 2.5 times ULN; aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 3 times ULN.
    3. Renal: Serum creatinine ≤ 1.5 x ULN.
18. Resolution of all acute toxic effects of prior surgical procedures to grade ≤1 as determined by the NCI CTCAE v.5.0.

Exclusion criteria

Patients will be excluded from the study if they meet ANY of the following criteria:

1. Metastatic progression (M1, according to TNM staging system).
2. Substantial nodal involvement (N>2, according to TNM staging system).
3. Non-large tumor (T0-1, according to TNM staging system).
4. Bilateral breast carcinoma.
5. Inflammatory carcinoma (T4d, according to TNM staging system).
6. Patient with multicentric or multifocal (more than 2 lesions) breast cancer.
7. Excisional biopsy of the primary tumor.
8. Known hypersensitivity to any palbociclib excipients.
9. Known hypersensitivity to any letrozole excipients.
10. Patients unable to swallow tablets.
11. Patients have a concurrent malignancy or malignancy within five years of study enrollment with the exception of carcinoma in situ of the cervix, non-melanoma skin carcinoma, or stage I uterine cancer. For other cancers considered to have a low risk of recurrence, discussion with the Medical Monitor is required.
12. Previous radiotherapy on the ipsilateral chest wall for the treatment of any other malignancy.
13. Major surgery (defined as requiring general anesthesia) or significant traumatic injury within four weeks of start of study treatment, or patients who have not recovered from the side effects of any major surgery, or patients that may require major surgery during the course of the study.
14. Have a serious concomitant systemic disorder (i.e., active infection including HIV, or cardiac disease) incompatible with the study (at the discretion of investigator).
15. Patients with an active bleeding diathesis, previous history of bleeding diathesis, or anti-coagulation treatment (the use of low molecular weight heparin is allowed as soon as it is used as prophylaxis intention).
16. History of malabsorption syndrome or other condition that would interfere with enteral absorption.
17. Chronic daily treatment with corticosteroids with a dose of ≥ 10mg/day methylprednisolone equivalent (excluding inhaled steroids).
18. QTc interval > 480 msec on basal assessments, personal history of long or short QT syndrome, Brugada syndrome or known history of QTc prolongation, or Torsade de Pointes (TdP).
19. Uncontrolled electrolyte disorders that can compound the effects of a QTc-prolonging drug (i.e., hypocalcemia, hypokalemia, or hypomagnesemia).
20. Participation in the treatment phase of an interventional trial within 30 days prior to study treatment start.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Pre and post menopausal females
Enrollment: 66 (Actual)
Dates: Start 2019-05-07 (Actual); Primary Completion 2019-07-30 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Difference on Recurrence Score between pre and post-treatment (molecular results) | 6 months
  To explore after 6 months of treatment the ability of palbociclib in combination with letro-zole to induce global molecular changes measured by either the Oncotype DX Breast Recurrence Score® (the "Assay") test result at surgery (post-treatment Recurrence Score® (RS) result), or pathological Complete Response (pCR) in patients with aggres-sive luminal tumors (pre-treatment RS result 18-25 or 26-100, and Ki67>20).

SECONDARY OUTCOMES:
Molecular changes | 6 months
  Concordance rate among post-treatment RS result and residual cancer burden (RCB), Ki67, and preoperative endocrine prognostic index (PEPI) score
Molecular induction | 6 months of treatment
  To explore the ability of palbociclib in combination with letrozole to induce global mo-lecular reduction measured by either the post-treatment RS result, and/or Residual Cancer Burden (RCB), and/or Ki67 in patients with aggressive luminal tumors (pre-treatment RS result 18-25 or 26-100 and Ki67>20) after 6 months of treatment.
Global molecular reduction | 6 months of treatment
  To verify the ability of palbociclib in combination with letrozole to induce global mo-lecular changes (measured as either post-treatment RS≤25 or RCB score of 0-I) in >35% of patients in cohort B with pre-treatment RS 26-100;
increase RS result | 6 months of treatment
  To verify the ability of palbociclib in combination with letrozole to induce changes in RS result (measured as post-treatment RS 26-100) in <3% of patients in cohort A with pre-treatment RS 18-25;
Evaluate the concordance rate between the RCB score (0- I vs. II-III) and the post-treatment RS result in both cohorts of patients after treatment with palbociclib in com-bination with letrozole; | 6 months of treatment
  To evaluate the concordance rate between the RCB score (0- I vs. II-III) and the post-treatment RS result in both cohorts of patients after treatment with palbociclib in com-bination with letrozole;
Evaluate the concordance rate between the pCR and the post-treatment RS re-sult in both cohorts of patients after treatment with palbociclib in combination with letro-zole; | 6 month of treatment
  To evaluate the concordance rate between the pCR and the post-treatment RS re-sult in both cohorts of patients after treatment with palbociclib in combination with letro-zole;
Changes in RS | 6 month of treatment
  To determine the change in RS result as measured by median absolute value or median percentage after 6 months of treatment: from pre-treatment RS 18-25 to post-treatment RS 0-17 for patients in cohort A and from pre-treatment RS 26-100 to post-treatment RS≤25 for patients in cohort B.

OTHER OUTCOMES:
overall repsonse | 6 month of treatment
  To determine the Overall Response Rate (ORR) of patients treated with palbociclib in combination with letrozole.
duration of response | 6 month of treatment
  To evaluate the Duration of Response (DoR) of palbociclib in combination with letrozole.
Time to response | 6 month of treatment
  To evaluate the Time to Response (TTR) of palbociclib in combination with letrozole.
Clinical benefit | 6 month of treatment
  To assess the Clinical Benefit Rate (CBR) of palbociclib in combination with letrozole.
Evaluate the Maximum Tumor Shrinkage of palbociclib in combination with letrozole | 6 month of treatment
  To evaluate the Maximum Tumor Shrinkage of palbociclib in combination with letrozole
Safety and tolerability of the combination Letrozole plus Palbociclib | 6 month of treatment
  To assess the safety and tolerability of palbociclib in combination with letrozole. "Number of participants with treatment-related adverse events as assessed by CTCAE v4.0".

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Llombart, PdH, Principal Investigator — MedSIR
Locations (18):
- Portugal (3):
  - Hospital da Luz, Lisbon
  - Hospital Fernando Fonseca, Lisbon
  - Portuguese Institute of Oncology of Oporto, Porto
- Spain (15):
  - ICO Badalona, Badalona, Barcelona
  - ICO l'Hospitalet, L'Hospitalet de Llobregat, Barcelona
  - Hospital de Jaén, Jaén, Jaén
  - Complejo Hospitalario Universitario A Coruña (CHUAC), A Coruña
  - H. Vall Hebrón, Barcelona
  - Hospital del Mar, Barcelona
  - Hospital Reina Sofia, Córdoba
  - Onkologikoa, Donostia / San Sebastian
  - Hospital Arnau de Vilanova, Lleida
  - Hospital Ramón y Cajal, Madrid
  - Hospital Universitario Virgen del Rocío, Seville
  - Instituto Valenciano de Oncologia, Valencia
  - Hospital Arnau de Vilanova de Valencia, Valencia
  - Hospital Clinico Universitario de Valencia, Valencia
  - Hospital Miguel Servet, Zaragoza

IPD SHARING:
Plan to Share IPD: Yes
20 hospital will participate at this trial: 17 sites at Spain and 3 at Portugal
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The trial separate 2 stage: Stage I it will be radomized 26 patients (20 Sites) from January 2019 to June2019 and Stage II: 40 patients (25 sites) from February 2020 to July 2020.
Access Criteria: patient should be randomized od Data base of hospitals